CLINICAL TRIAL: NCT03079024
Title: Minnesota Community-Based Cognitive Training in Early Psychosis
Acronym: Mini-COTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSYCH-2017-25503
Record Dates: First submitted 2017-02-09; First posted 2017-03-14 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia; Psychosis; Schizoaffective Disorder; Schizophreniform Disorders; Psychosis NOS; Depression Psychotic Feature; Bipolar Disorder With Psychotic Features; Unspecified Psychosis
Keywords: Cognitive Training; First Episode Psychosis; Recent Onset Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Targeted Cognitive Training (TCT) (Experimental): Neuroadaptive Cognitive Training
  Interventions: Device: Targeted Cognitive Training; Other: Coordinated Specialty Care for First Episode Psychosis
- General Cognitive Exercises (GCE) (Experimental): Neuroadaptive cognitive training
  Interventions: Device: General Cognitive Exercises; Other: Coordinated Specialty Care for First Episode Psychosis
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual
  Interventions: Other: Coordinated Specialty Care for First Episode Psychosis

INTERVENTIONS:
Device: Targeted Cognitive Training — 1. Auditory Training Module (20 hours): exercises designed to improve speed and accuracy of auditory processing while engaging working memory and cognitive control. Exercises adjust difficulty level to maintain an ~80% correct performance. Exercises contain stimuli spanning the acoustic organization of speech. In the initial stages, stimuli exaggerate the rapid temporal transitions by increasing amplitude and stretching in time. The exaggeration is gradually removed so that by the end, all stimuli have characteristics representative of real-world speech.
  2. Social Cognition Module (10 hours): exercises designed to improve core deficits of social cognition in psychosis. Exercises apply principles of implicit learning to restore capacity to process and utilize socially-relevant information, and includes training to improve perception of affect (visual/vocal) and social cues (faces, gazes, social situations), theory of mind, self-referential style, emotion labeling and working memory.
  Arms: Targeted Cognitive Training (TCT)
Device: General Cognitive Exercises — The GCE will focus on executive dysfunction, as this domain is a significant, functionally important area of deficit in schizophrenia and has been the target of many previous studies. We will train this domain using a suite of engaging, adaptive web-based exercises that target executive function, intelligence, and spatial navigation developed by Posit Science. The exercises will be provide engaging, adaptive training as described in the Targeted Cognitive Training.
  Arms: General Cognitive Exercises (GCE)
Other: Coordinated Specialty Care for First Episode Psychosis — Individuals in this study are receiving care from a coordinated specialty care clinic (CSC) for first episode psychosis. These clinics are following the NAVIGATE treatment model for early psychosis.

SUMMARY:
The purpose of this study is to determine whether cognitive training exercises can improve cognitive functioning in young patients with recent-onset psychosis who are being treated in community mental health settings using the NAVIGATE model. The investigators will examine the effects of web-based cognitive training exercises delivered on iPads. Participants will be randomized to one of three conditions, and will be assessed at Baseline, Post-Intervention, and 6 Month Follow Up on measures of clinical, neurocognitive, and functional status.

DETAILED DESCRIPTION:
The purpose of this study is to perform a double-blind randomized controlled trial (RCT) in young patients with First Episode Psychosis (FEP) to target improvement in cognitive functioning within real-world treatment settings. This study will be performed in the University of Minnesota Department of Psychiatry; patients will be recruited from local community based mental health care settings that implement a NAVIGATE model for FEP.

All participants will undergo baseline assessment in measures of clinical, neurocognitive, and functional status prior to randomization. Participants will be equally randomized to one of three groups: Targeted Cognitive Training (TCT); General Cognitive Exercises (GCE); or Treatment as Usual (TAU). Participants assigned to a cognitive training group will be loaned an iPad to complete study training at home. They will complete 60 minutes of training 5 times a week over the course of 6 weeks for a total of 30 hours of training. Participants will be allowed up to 12 weeks to complete the full 30 hours. Participants will return after 30 hours of training or 12 weeks, whichever comes first, for Post-Intervention Assessments. Then participants will enter a no-contact follow up period, until it is time for their 6 Month Follow Up assessment.

Specific Aims:

1. Perform a double-blind RCT of web-based, portable computerized cognitive training in young individuals with recent onset psychosis receiving treatment within the University of Minnesota, Department of Psychiatry's First Episode Psychosis Program or other state clinics utilizing the NAVIGATE treatment model.
2. Compare the clinical and cognitive effects of neural system-informed TCT that focuses explicitly and specifically on distributed neural system efficiency in auditory/verbal and social cognitive domains, vs. more non-specific GCE designed to enhance executive functioning and problem-solving, vs. TAU. Determine the durability of these effects and their relationship to functional outcome over a 6 month period.
3. As a secondary aim, investigate the feasibility, tolerability, and acceptability of the intervention by service providers, clients, and caregivers in these real-world treatment centers.

Hypotheses to be tested:

1. TCT subjects will show significantly greater gains in general cognition, verbal learning/memory, and social cognition compared to GCE and TAU subjects. These gains in the TCT group will be sustained at 6-month follow-up.
2. GCE subjects will show improvement in problem-solving and global cognition compared to TAU subjects. At 6 month follow-up, GCE subjects will show lower gains in global cognition and verbal learning/memory than TCT subjects.
3. Gains in general cognition and processing speed, and in social cognition in TCT subjects will correlate with improvements on 6-month measures of occupational and social functioning, respectively, as well as internalized stigma. These associations will be significantly greater in TCT subjects vs. GCE or TAU subjects.
4. Symptom ratings will show improvement in all subject groups at 6 months, with no significant between-group differences.
5. At least 70% of randomized clients will complete >20 hours of training in the TCT and GCE arms.
6. Participants and clinicians will rate the TCT and GCE interventions as equally feasible, tolerable, and acceptable.

Participants from this study will also be recruited to participate in an adjunct protocol conducted by Dr. Sophia Vinogradov, titled "Is cognitive training neuroprotective in early psychosis?" NCT03049800.

Data from this project will be analysed with a sister protocol conducted by Dr. Rachel Loewy at the University of California San Francisco, titled "Community-Based Cognitive Training in Early Schizophrenia (COTES)," NCT01973270.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, major depressive disorder with psychotic features, bipolar disorder with psychotic features, psychosis disorder not otherwise specified, or unspecified schizophrenia spectrum disorder, and started receiving treatment services at a First Episode Psychosis Program within the last two years
* Good general physical health
* Aged between 16 and 35 years (inclusive)
* Fluent in spoken and written English
* No neurological disorder (diagnosis of Autism Spectrum Disorder is allowed)
* Achieved clinical stability, defined as outpatient status for at least one month prior to study participation, stable doses of psychiatric medications for at least one month prior to study participation
* Women who are pregnant or breastfeeding may participate in this study.

Exclusion Criteria:

* Unable to provide informed consent
* Participated in significant cognitive training programs within the last three years
* Clinically significant substance abuse that is impeding the subject's ability to participate fully during recruitment, assessment, or training (is unable to remain sober for assessments and training).
* Prescribed >0.5mg daily benztropine (Congentin), >25mg daily diphenhydramine, or high doses of clozapine (>500 mg po qd) or olanzapine (to be determined on a case by case basis).
* Active suicidal ideation at screening or baseline, or previous intent to act on suicidal ideation with a specific plan, preparatory acts, or an actual suicide attempt within the last 6 months, as indicated by the C-SSRS

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2022-03-26 (Actual); Study Completion 2022-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota Department of Psychiatry
Locations (1):
- University of Minnesota, Dept of Psychiatry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
All assessment and training data and supporting information may be made available to collaborators upon request. Collaborators will need to enter into proper agreements with the PI and Institution before access is granted.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Study data will be available for sharing one year after the completion of the project.
Access Criteria: Interested collaborators may contact the PI directly to request access to the study data. Collaborators will need to enter into Data Use Agreements with the PI and Institution, and limitations may be made on how data is shared (e.g., within a data shelter).

RESULTS

PARTICIPANT FLOW:
Groups:
- Targeted Cognitive Training (TCT): Neuroadaptive Cognitive Training
  Targeted Cognitive Training: 1. Auditory Training Module (20 hours): exercises designed to improve speed and accuracy of auditory processing while engaging working memory and cognitive control. Exercises adjust difficulty level to maintain an ~80% correct performance. Exercises contain stimuli spanning the acoustic organization of speech. In the initial stages, stimuli exaggerate the rapid temporal transitions by increasing amplitude and stretching in time. The exaggeration is gradually removed so that by the end, all stimuli have characteristics representative of real-world speech.
  2. Social Cognition Module (10 hours): exercises designed to improve core deficits of social cognition in psychosis. Exercises apply principles of implicit learning to restore capacity to process and utilize socially-relevant information, and includes training to improve perception of affect (visual/vocal) and social cues (faces, gazes, social situations), theory of mind, self-referential style, emotion labeling and working memory.
  Coordinated Specialty Care for First Episode Psychosis: Individuals in this study are receiving care from a coordinated specialty care clinic (CSC) for first episode psychosis. These clinics are following the NAVIGATE treatment model for early psychosis.
Period: Overall Study
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Started | 16 | 17 | 12
Completed | 13 | 14 | 9
Not Completed | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 16 | 17 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.88 (3.22) | 20.59 (4.37) | 22 (3.38) | 21.07 (3.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 8
  Male | 13 | 16 | 8 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 6
  White | 10 | 12 | 7 | 29
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Speed of Processing From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: A composite T-score of:
  1. Symbol Coding from the Brief Assessment of Cognition in Schizophrenia (BACS): Symbol Coding. Timed paper-and-pencil test in which respondent uses a key to write digits that correspond to nonsense symbols.
  2. Category Fluency: Animal Naming: Oral test in which respondent names as many animals as she/he can in 1 minute.
  3. Trail Making Test: Part A: Timed paper-and-pencil test in which respondent draws a line to connect consecutively numbered circles placed irregularly on a sheet of paper. The composite T-score is the average T-score across the 3 measures. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T- score of 50 indicates the population mean (average) with a standard deviation of
  10.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 15 | 11
T-score | 41.75 (8.75) | 41.2 (12.74) | 24.82 (14.5)

2. Primary Outcome: Speed of Processing From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 7
T-score | 49.5 (13.96) | 39.22 (12.43) | 41.57 (14.01)

3. Primary Outcome: Speed of Processing From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 1
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 2
T-score | 48.4 (13.13) | 40.56 (10.62) | 51.5 (16.26)

4. Primary Outcome: Attention From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Continuous Performance Test-Identical Pairs (CPT-IP): A computer- administered measure of sustained attention in which respondent presses a response button to consecutive matching numbers. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 15 | 10
T-score | 37.38 (10.83) | 35.2 (9.17) | 34.5 (8.92)

5. Primary Outcome: Attention From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 4
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 6
T-score | 42.4 (9.52) | 36.89 (11.17) | 41.67 (7.37)

6. Primary Outcome: Attention From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 4
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 8 | 2
T-score | 40.6 (11.3) | 37.5 (8.91) | 39.5 (3.54)

7. Primary Outcome: Working Memory From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Verbal and Visual Working Memory: A composite score of the Letter- Number Span test and the Spatial Span test from the Wechsler Memory Scale®-3rd Ed. (WMS®-III). Letter-Number Span: An orally administered test in which respondent mentally reorders strings of number and letters and repeats them to administrator. Spatial Span: Using a board on which 10 cubes are irregularly spaced, respondent taps cubes in same (or reverse) sequence as test administrator. The composite T-score is the average T-score across the 2 measures. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: Basline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 17 | 12
T-score | 44.13 (10.4) | 43.88 (11.11) | 39.17 (8.5)

8. Primary Outcome: Working Memory From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 7
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 9
T-score | 43.5 (12.06) | 43.29 (12.64) | 43.8 (4.49)

9. Primary Outcome: Working Memory From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 7
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11 | 5
T-score | 43.75 (11.05) | 41.91 (11.92) | 43.8 (4.49)

10. Primary Outcome: Verbal Learning From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Hopkins Verbal Learning Test-Revised (HVLT-R): An orally
  administered test in which a list of 12 words from three taxonomic categories is presented and the respondent is asked to recall as many as possible after each of three learning trials. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 17 | 12
T-score | 43.06 (9.17) | 42.71 (9.36) | 36.83 (7.85)

11. Primary Outcome: Verbal Learning From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 10
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 9
T-score | 42.6 (7.26) | 43.57 (9.08) | 40.22 (8.57)

12. Primary Outcome: Verbal Learning From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 10
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11 | 5
T-score | 43.67 (10.25) | 42.73 (8.38) | 46.2 (14.32)

13. Primary Outcome: Visual Learning From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Brief Visuospatial Memory Test-Revised (BVMT-RTM): A test that involves reproducing six geometric figures from memory. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 15 | 10
T-score | 43.63 (12.25) | 42.53 (6.82) | 36.6 (8.66)

14. Primary Outcome: Visual Learning From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 13
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 7
T-score | 42.7 (13.65) | 41.33 (8.43) | 43.14 (10.99)

15. Primary Outcome: Visual Learning From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 13
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 2
T-score | 44.4 (14.34) | 42.89 (7.41) | 47 (15.56)

16. Primary Outcome: Problem Solving From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Neuropsychological Assessment Battery® (NAB®): Mazes: Seven timed paper-and-pencil mazes of increasing difficulty that measure foresight and planning. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 15 | 10
T-score | 40.06 (10.81) | 38.67 (8.8) | 36 (13.93)

17. Primary Outcome: Problem Solving From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 16
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 7
T-score | 46.4 (11.34) | 42 (9.8) | 39 (11.37)

18. Primary Outcome: Problem Solving From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 16
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 2
T-score | 49.3 (9.92) | 42.11 (10.01) | 44.5 (20.51)

19. Primary Outcome: Social Cognition From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: Mayer-Salovey-Caruso Emotional Intelligence Test(MSCEIT™ ): Managing Emotions: Paper-and-pencil multiple-choice test that assesses how people manage their emotions. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 17 | 12
T-score | 42.75 (10.27) | 44.24 (9.83) | 45.58 (11.89)

20. Primary Outcome: Social Cognition From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 19
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 9
T-score | 46.4 (12.19) | 41.93 (9.57) | 47.44 (11.68)

21. Primary Outcome: Social Cognition From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 19
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11 | 5
T-score | 43.75 (9.21) | 44.73 (7.86) | 52.6 (12.18)

22. Primary Outcome: Global Cognition From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: A composite score of the 7 scores listed above: Speed of Processing, Attention, Working Memory, Verbal Learning, Visual Learning, Problem Solving, and Social Cognition. The composite T-score is the average T-score across the 7 measures. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 15 | 10
T-score | 36.75 (11.41) | 35.4 (11.56) | 29.6 (10.59)

23. Primary Outcome: Global Cognition From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 22
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 6
T-score | 41.5 (12.96) | 33.78 (11.99) | 37.5 (10.95)

24. Primary Outcome: Global Cognition From the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: as for outcome 22
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 8 | 2
T-score | 41.6 (14.82) | 39.63 (8.37) | 45 (19.8)

25. Primary Outcome: Emotion Recognition From the University of Pennsylvania Computerized Neurobehavioral Test Battery
Description: Emotion Recognition: Participants are shown a series of 40 faces, one at a time, and asked to determine what emotion the face is showing for each trial. There are 5 answer choices: happy, sad, anger, fear and no emotion. Scores (i.e. correct responses) range from 0-40 with higher scores corresponding to better performance.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Total correct responses
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 14 | 10
Total correct responses | 32.56 (4.05) | 31.50 (3.7) | 32.5 (2.07)

26. Primary Outcome: Emotional Prosody Identification From the University of Pennsylvania Computerized Neurobehavioral Test Battery Neurobehavioral Test Battery
Description: Emotional Prosody Identification: Participants are presented a series of 80 audio clips played one at a time, and asked to determine what emotion the audio clip portrayed. There are 5 answer choices: Happy, Sad, Anger, Fearful and No Emotion. Scores (i.e. correct responses) range from 0-80 with higher scores corresponding to better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Total correct responses
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 14 | 10
Total correct responses | 37.94 (6.41) | 39.64 (8.83) | 37.8 (11.3)

27. Primary Outcome: Emotional Prosody Identification From the University of Pennsylvania Computerized Neurobehavioral Test Battery
Description: as for outcome 26
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Total correct responses
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 9 | 6
Total correct responses | 44.63 (3.96) | 40.89 (6.85) | 41.67 (5.2)

28. Primary Outcome: Emotion Recognition From the University of Pennsylvania Computerized Neurobehavioral Test Battery
Description: as for outcome 25
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Total correct responses
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 7 | 6
Total correct responses | 34.88 (3.32) | 32.29 (2.75) | 33.67 (3.33)

29. Primary Outcome: Emotion Recognition From the University of Pennsylvania Computerized Neurobehavioral Test Battery
Description: as for outcome 25
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Total correct responses
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 7 | 2
Total correct responses | 34.9 (1.79) | 32.71 (2.21) | 33.5 (2.12)

30. Primary Outcome: Emotional Prosody Identification From the University of Pennsylvania Computerized Neurobehavioral Test Battery
Description: as for outcome 26
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Total correct responses
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 7 | 2
Total correct responses | 41.1 (6.23) | 43.29 (6.24) | 41 (1.41)

31. Primary Outcome: Faux Pas Test Theory of Mind
Description: Faux Pas Test: Brief stories are read to the participant, and the participant is asked if someone in the story made a faux pas. This test assesses the ability to infer other peoples' mental states, thoughts and feelings. Scores (i.e. percent correct) range from 0-100% with higher scores corresponding to better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 11 | 15 | 12
Percent | 83.79 (6.06) | 89.33 (7.99) | 82.78 (15.08)

32. Primary Outcome: Faux Pas Test Theory of Mind
Description: as for outcome 31
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 8 | 14 | 9
Percent | 79.38 (17.3) | 91.24 (6.9) | 81.85 (13.27)

33. Primary Outcome: Faux Pas Test Theory of Mind
Description: as for outcome 31
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11 | 5
Percent | 82.36 (13.23) | 89.39 (12) | 91.67 (5.89)

34. Primary Outcome: Quality of Life Scale-Abbreviated (Functioning)
Description: Functioning: This measure assesses quality of life using subjective questions regarding life satisfaction and objective indicators of social and occupational functioning. Participants are asked questions about social and occupational functioning and intrapsychic foundations (e.g. motivation, sense of purpose, curiosity). The assessor provides ratings on a scale of 0-6 (e.g. absent to adequate). A mean item score is computed as the average rating across all items, with higher mean item scores corresponding to better functioning.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 17 | 12
Mean item score | 3.69 (1.25) | 3.75 (1.09) | 3.72 (1.1)

35. Primary Outcome: Quality of Life Scale-Abbreviated (Functioning)
Description: as for outcome 34
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 8
Mean item score | 4.6 (1.06) | 3.95 (1.1) | 4.49 (0.79)

36. Primary Outcome: Quality of Life Scale-Abbreviated (Functioning)
Description: as for outcome 34
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: Mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11 | 5
Mean item score | 4.25 (1.02) | 3.66 (1.29) | 4.67 (0.46)

37. Primary Outcome: Auditory Processing Speed From the Posit Science Sound Sweeps Assessment
Description: Auditory Processing Speed: In Sound Sweeps, participants listen to frequency sweeps-sounds that begin low and rise upward or begin high and fall downward-and identify whether they go up ("weep") or down ("woop"). The sweeps become progressively faster and are separated by shorter interstimulus intervals. The outcome is the threshold reached by the participant which is the fastest interstimulus interval (in milliseconds) at which the participant correctly performed. Scores ranged from 24-1000 milliseconds with lower scores indicating better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 7 | 9 | 11
Milliseconds | 275.43 (357.14) | 124.33 (70.87) | 181.64 (169.41)

38. Primary Outcome: Auditory Processing Speed From the Posit Science Sound Sweeps Assessment
Description: as for outcome 37
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 4 | 10 | 6
Milliseconds | 73 (21.56) | 76.5 (39.78) | 87.67 (40.71)

39. Primary Outcome: Auditory Processing Speed From the Posit Science Sound Sweeps Assessment
Description: as for outcome 37
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 9 | 9 | 5
Milliseconds | 166.44 (165.09) | 103.67 (59.55) | 99.2 (89.4)

40. Primary Outcome: Temporal Experience of Pleasures (TEPS):Reward Sensitivity--Anticipatory Pleasure
Description: Reward Sensitivity--Anticipatory Pleasure: This measure assesses pleasure experienced in anticipation of something and consists of 10 items. An example item is: "When something exciting is coming up in my life, I really look forward to it." Participants rate how true the statement is for them on a scale of 1 (very false for me) to 6 (very true for me). A mean item score is computed as the average rating across all items, with higher mean item scores corresponding to greater anticipatory pleasure.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 15 | 17 | 12
mean item score | 4.08 (0.66) | 4.1 (0.72) | 4.01 (0.6)

41. Primary Outcome: Temporal Experience of Pleasures (TEPS):Reward Sensitivity--Anticipatory Pleasure
Description: as for outcome 40
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 8
mean item score | 3.87 (0.71) | 4.09 (0.62) | 4.93 (0.7)

42. Primary Outcome: Temporal Experience of Pleasures (TEPS):Reward Sensitivity--Anticipatory Pleasure
Description: as for outcome 40
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 11 | 5
mean item score | 4.25 (0.79) | 4.17 (0.67) | 4.42 (0.53)

43. Primary Outcome: Temporal Experience of Pleasures (TEPS): Reward Sensitivity--Consummatory Pleasure
Description: Reward Sensitivity--Consummatory Pleasure: This measure assesses pleasure experienced in the moment and consists of 8 items. An example item is: "The smell of freshly cut grass is enjoyable to me." Participants rate how true the statement is for them on a scale of 1 (very false for me) to 6 (very true for me). A mean item score is computed as the average rating across all items, with higher mean item scores corresponding to greater consummatory pleasure.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Mean Item Score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 17 | 12
Mean Item Score | 4.66 (0.72) | 4.26 (1.07) | 4.47 (0.54)

44. Primary Outcome: Temporal Experience of Pleasures (TEPS): Reward Sensitivity--Consummatory Pleasure
Description: as for outcome 43
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Mean Item Score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 8
Mean Item Score | 4.98 (0.55) | 4.7 (0.56) | 4.86 (0.47)

45. Primary Outcome: Temporal Experience of Pleasures (TEPS): Reward Sensitivity--Consummatory Pleasure
Description: as for outcome 43
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: Mean Item Score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 11 | 5
Mean Item Score | 4.89 (0.66) | 4.78 (0.66) | 4.93 (0.56)

46. Primary Outcome: Verbal Memory: Delayed Recall From the Hopkins Verbal Learning Test-Revised Version (HVLT-R)
Description: Verbal Memory: Delayed Recall: An orally administered test in which a list of 12 words from three taxonomic categories is presented and the respondent is asked to recall as many as possible after a 25 minute delay. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 16 | 12
T-score | 42.55 (12.54) | 41.15 (13.06) | 32.61 (14.78)

47. Primary Outcome: Verbal Memory: Delayed Recall From the Hopkins Verbal Learning Test-Revised Version (HVLT-R)
Description: as for outcome 46
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 13 | 8
T-score | 40.69 (14.18) | 35.73 (13.42) | 37.61 (19.51)

48. Primary Outcome: Verbal Memory: Delayed Recall From the Hopkins Verbal Learning Test-Revised Version (HVLT-R)
Description: as for outcome 46
Time Frame: 6months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11 | 5
T-score | 41.32 (13.87) | 36.31 (20.57) | 38.39 (22.17)

49. Primary Outcome: Visual Memory: Delayed Recall From the Brief Visuospatial Memory Test-Revised Version (BVMT-R)
Description: Visual Memory: Delayed Recall: A test that involves reproducing six geometric
  figures from memory after a 25 minute delay. T-scores range from 0-100, with higher T-scores corresponding to better performance. A T-score of 50 indicates the population mean (average) with a standard deviation of 10.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 15 | 10
T-score | 46.48 (10.85) | 46.86 (13.72) | 43.09 (14.62)

50. Secondary Outcome: UCSF Performance-Based Skills Assessment (UPSA): Functional Capacity
Description: Functional Capacity: This measure assesses how well everyday tasks are performed in two areas of functioning: communication (e.g. making an emergency call, calling a doctor to reschedule an appointment) and finances (e.g. counting change, reading a utility bill). Scaled scores range from 0-100 with higher scores indicating better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 15 | 10
Total score | 73.58 (12.4) | 73.33 (16.48) | 69.14 (9.71)

51. Secondary Outcome: UCSF Performance-Based Skills Assessment (UPSA): Functional Capacity
Description: as for outcome 50
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 7
Total score | 76.31 (9.24) | 61.05 (13.63) | 70.92 (14.66)

52. Secondary Outcome: UCSF Performance-Based Skills Assessment (UPSA): Functional Capacity
Description: as for outcome 50
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 11 | 9 | 5
Total score | 67.86 (25.74) | 69.42 (6.61) | 30.1 (41.4)

53. Secondary Outcome: Social Functioning Scale
Description: Social Functioning: This measure assesses social skills and functioning in 7 domains: Withdrawal, Interaction, Pro-Social, Recreation, Independence- Performance, Independence-Competence, and Occupational. A mean domain score was calculated as the average across all domains. Scaled scores range from 55-145 with higher scores indicating better functioning.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: subscale score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 17 | 12
subscale score | 106.45 (8.09) | 106.73 (9.2) | 107.15 (7.71)

54. Secondary Outcome: Social Functioning Scale
Description: as for outcome 53
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: subscale score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 8
subscale score | 113.33 (5.09) | 107 (8.49) | 117.05 (5.89)

55. Secondary Outcome: Social Functioning Scale
Description: as for outcome 53
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: subscale score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 12 | 11 | 5
subscale score | 112.43 (8.06) | 107.58 (10.47) | 121.09 (5.05)

56. Secondary Outcome: Internalized Stigma of Mental Illness (ISMI)
Description: This measure assesses internalized stigma which occurs when a person adopts stigmatizing assumptions and stereotypes about mental illness. Participants rate 10 statements on a scale of 1 (strongly disagree) to 4 (strongly agree). A mean item score is computed as the average rating across all items, with higher mean item scores corresponding to greater internalized stigma.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 16 | 17 | 12
Mean item score | 1.76 (0.44) | 2.11 (0.44) | 2.04 (0.47)

57. Secondary Outcome: Internalized Stigma of Mental Illness (ISMI)
Description: as for outcome 56
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 14 | 8
Mean item score | 1.79 (0.38) | 1.89 (0.33) | 1.69 (0.45)

58. Secondary Outcome: Internalized Stigma of Mental Illness (ISMI)
Description: as for outcome 56
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: Mean item score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 10 | 5
Mean item score | 1.74 (0.42) | 2.14 (0.32) | 1.46 (0.3)

59. Primary Outcome: Visual Memory: Delayed Recall From the Brief Visuospatial Memory Test-Revised Version (BVMT-R)
Description: as for outcome 49
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 7
T-score | 46.62 (14.4) | 43.64 (8.66) | 46.16 (12.8)

60. Primary Outcome: Visual Memory: Delayed Recall From the Brief Visuospatial Memory Test-Revised Version (BVMT-R)
Description: as for outcome 49
Time Frame: 6 months followup
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
Number analyzed (Participants) | 10 | 9 | 2
T-score | 48.67 (14.37) | 48.16 (9.22) | 46.89 (9.56)

ADVERSE EVENTS:
Time Frame: Participants were randomized to 30 hours of TCT or GCE training or 12 weeks (whichever came first), or 12 weeks of TAU and completed baseline, post-intervention and 6 month follow-up assessments.
Arm/Group | Targeted Cognitive Training (TCT) | General Cognitive Exercises (GCE) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/16 | 3/17 | 1/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Cognitive Training (TCT) (N=16) | General Cognitive Exercises (GCE) (N=17) | Treatment as Usual (TAU) (N=12)
Hospitialization unrelated to study procedures. (General disorders) | 2 (4) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Missing data: This study was conducted from 2017-2022. During the COVID-19 shutdown, we continued the study and shifted to all remote procedures, however several measures could not be administered remotely. 2. The BACS Tower of London was not administered to reduce participant burden, and since Reasoning and Problem Solving was already captured by the MATRICS battery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT03079024/Prot_SAP_000.pdf